CLINICAL TRIAL: NCT05250986
Title: Comparison of Visual Acuity Performed in Office Versus In Residence
Acronym: VA IR vs IO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gobiquity Mobile Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-001
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: GoCheck Kids (iOS) — Visual Acuity method is used to measure of the sharpness or clearness of vision.
  Device: GoCheck Visual Acuity in Office (Windows) Photorefraction method is used to screen amblyopia risk factors.
Device: GoCheck Kids (Windows) — Visual Acuity method is used to measure of the sharpness or clearness of vision.
Device: GoCheck at Home (iOS) — Visual Acuity method is used to measure of the sharpness or clearness of vision.
Device: GoCheck at Home (Windows) — Visual Acuity method is used to measure of the sharpness or clearness of vision.

SUMMARY:
GoCheck has developed and deployed a home-based visual acuity test that may be used in-office or in residence. The test methodology utilizes modified ATS and ETDRS protocols with Sloan optotypes, crowding bars and sophisticated algorithms. The objective of this study is to determine if the results of the GoCheck visual acuity test performed in an office setting correlate to the same testing when implemented in the residence

DETAILED DESCRIPTION:
To address the increasing needs for remote patient assessment, GoCheck has developed and deployed a home-based visual acuity test that may be used in-office or in residence, to meet the changing needs of providers visit time allocation, as well as presenting a standardized form of visual acuity centered around clinically-validated approaches.

The test methodology utilizes modified ETDRS design features with HOTV or Sloan optotypes (based on age), crowding bars, and displays 3 optotypes at a time (arranged vertically) to accommodate smaller screen sizes, but still significantly shortens testing time as opposed to displaying only a single optotype at a time.

The application may be used to screen children old enough to comprehend the test, typically around age 4 through adulthood, during their primary care, or school-based visits, and now, in the home. The purpose of home vision testing is to provide actionable insights into the status of an individual's vision without the need for an in-office visit. The testing results will be able to used by the physician to help determine if additional interventions are necessary.

The objective of this study is to determine if the results of the GoCheck visual acuity test performed in an office setting correlate to the same testing when implemented in the residence.

ELIGIBILITY:
Inclusion Criteria:

1. Ages four (4) to twenty(20) years, inclusive
2. Corrected visual acuity range of 20/16 to 20/100
3. Manifest or cycloplegic refraction within prior six (6) months
4. Ability to comprehend and complete the VA test with age appropriate optotypes

Exclusion Criteria:

1. No access to smartphone
2. Inability to read, write, and/or understand English
3. Inability to provide written informed consent or have consent conferred on patient's behalf
4. Subjects from populations otherwise deemed ineligible/unable to provide informed consent and/or participate in studies (detention, correction, rehabilitation, psychiatric residents, etc.)
5. Current pregnancy
6. Any ocular pathology defect(s) except amblyopia, strabismus or refractive error or history of nystagmus.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: English-speaking individuals of any gender, aged four to twenty years, with recent refraction, able to comprehend and complete the visual acuity test with age appropriate optotypes.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2022-02-14 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of in-office visual acuity results to visual acuity results obtained in residence. | 10 Days
  correlation of visual acuity results obtained by trained personnel utilizing the GoCheck Kids Visual Acuity solution in an in-office clinical setting compared to the results obtained by individuals conducting the same visual acuity test in their residence.

SECONDARY OUTCOMES:
Accuracy of in residence visual acuity results to opthalmic visual acuity | 10 Days
  Accuracy of visual acuity results obtained in residence relative to standard ophthalmic visual acuity test.
Repeatability and Reproducibility of Visual Acuity in Residence | 7 Days
  The repeatability and reproducibility of results of visual acuity testing conducted in the residence within defined intervals

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, Study Chair — Oregon Health and Science University
Locations (4):
- United States (3):
  - Alaska Children's Eye & Strabismus, Anchorage, Alaska
  - Yale School of Medicine, Yale University, New Haven, Connecticut
  - Medical University of South Carolina-Storm Eye Institute, Charleston, South Carolina
- Stern Hospital, Haifa, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided